CLINICAL TRIAL: NCT04005105
Title: Acute Post-cardiac Surgery Renal Failure: Prevention Through Individualized Intensive Hemodynamic Management and Evaluation of Prognostic Biomarkers
Brief Title: Acute Post-cardiac Surgery Renal Failure: Prevention Through Individualized Intensive Hemodynamic Management
Acronym: PrevHemAKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Hospital Sant Joan de Deu (Other)
Responsible Party: Principal Investigator, Esteban Poch, Head of the Department of Nephrology and Kidney Transplantation, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PrevHemAKI
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive management (Active Comparator): Baseline mean blood pressure (MAP) and central venous pressure (CVP) will be measured to calculate baseline mean perfusion pressure. Intra-surgical values of ± 25% basal MAP will be maintained and once in the ICU an algorithm corresponding to group
  1 based on cardiac index and MPP will be followed for 24 hours.
  Interventions: Behavioral: Intensive management
- Standard management (No Intervention): MAP during surgery will be maintained > 60 mmHg according to usual protocol. Once in ICU, during the first 24 hours an algorithm corresponding to group 2 based on cardiac index, MAP and CVP will be followed.

INTERVENTIONS:
Behavioral: Intensive management — Management based on premorbid MAP and MPP
  Arms: Intensive management

SUMMARY:
BACKGROUND: The incidence of acute kidney injury (AKI) in patients undergoing cardiac surgery can reach 35% and between 2 and 5% require kidney replacement therapy during the AKI episode. The development of AKI n this context is independently associated with higher long-term mortality (5-10 years). In addition, there is strong evidence that an episode of AKI in the hospital increases the risk of developing chronic kidney disease in the medium-long term. On the other hand, once AKI has been recovered according to creatinine values, there are no established biomarkers to predict patients at risk of progression to chronic kidney disease, which will allow us to increase nephroprotection and surveillance measures in this group of patients.

STUDY DESIGN: Open-label randomized unicentric prospective study of patients undergoing valvular replacement heart surgery ± coronary bypass with acute kidney injury (AKI) risk >30% according to the Leicester Cardiosurgery scale. Patients will be randomized 1:1 in two groups: standard hemodynamic management or intensive hemodynamic management based on premorbid mean perfusion pressure (MPP). The interventional period will span from intra-operation until the first 24 hours postoperative. The incidence of AKI will be evaluated according to KDIGO criteria between 48 hours and 7 days after surgery. Patients will be followed for one year. Biomarkers of mitochondrial damage will be analyzed at various points during the follow-up to patients presenting AKI.

INTERVENTIONS:

A) Group 1/Intensive management: Intra-surgical values of ± 25% basal MAP will be maintained and once in the ICU an algorithm corresponding to group 1 based on cardiac index and ± 25% MPP will be followed for 24 hours.

B) Group 2/Standard management: MAP during surgery will be maintained > 60 mmHg according to usual protocol. Once in ICU, during the first 24 hours an algorithm corresponding to group 2 based on cardiac index, MAP and CVP will be followed.

Biomarkers of mitochondrial damage will be determined in urine in patients in both groups only in patients developing AKI according to KDIGO guidelines between 48h and 7 days.

EXPECTED RESULTS:A 50% reduction in the incidence of AKI in the intervention group compared to the control group is expected. At the same time, markers of mitochondrial damage are expected to be validated in our cohort as biomarkers of AKI progression and to investigate its usefulness as biomarkers of transition to Chronic kidney disease.

DETAILED DESCRIPTION:
BACKGROUND:

The incidence of acute kidney injury (AKI) in patients undergoing cardiac surgery can reach 35% and between 2 and 5% require kidney replacement therapy during the AKI episode. The development of AKI n this context is independently associated with higher long-term mortality (5-10 years). In addition, there is strong evidence that an episode of AKI in the hospital increases the risk of developing chronic kidney disease in the medium-long term. That is why the prevention of AKI is essential to reduce the morbidity that these patients suffer in the hospital and out-of-hospital environment. On the other hand, once AKI has been recovered according to creatinine values, there are no established biomarkers to predict patients at risk of progression to chronic kidney disease, which will allow us to increase nephroprotection and surveillance measures in this group of patients.

STUDY DESIGN:

Open-label randomized unicentric prospective study of patients undergoing valvular replacement heart surgery ± coronary bypass with acute kidney injury (AKI) risk >30% according to the Leicester Cardiosurgery scale. Patients will be randomized 1:1 in two groups: standard hemodynamic management or intensive hemodynamic management based on premorbid mean perfusion pressure (MPP). The interventional period will span from intra-operation until the first 24 hours postoperative. The incidence of AKI will be evaluated according to KDIGO criteria between 48 hours and 7 days after surgery. Patients will be followed for one year. Biomarkers of mitochondrial damage will be analyzed at various points during the follow-up to patients presenting AKI. Intention to treat population will be defined as patients who sign informed consent and undergo planned surgery.

INTERVENTIONS-ANALYSIS:

A) Group 1/Intensive management: Baseline mean blood pressure (MAP) and central venous pressure (CVP) will be measured to calculate baseline mean perfusion pressure (MPP). Intra-surgical values of ± 25% basal MAP will be maintained and once in the ICU an algorithm corresponding to group 1 based on cardiac index and ± 25% MPP will be followed for 24 hours.

B) Group 2/Standard management: MAP during surgery will be maintained > 60 mmHg according to usual protocol. Once in ICU, during the first 24 hours an algorithm corresponding to group 2 based on cardiac index, MAP and CVP will be followed. Biomarkers of mitochondrial damage will be determined in urine in patients in both groups only in patients developing AKI according to KDIGO guidelines between 48h and 7 days. The following variables will be assessed in both groups: accumulated fluid balance in first 24 hours, ICU /hospitalization length of stay, days with vasoactive support, MAKE (Major Adverse Kidney Events: mortality, need for renal replacement therapy, persistent renal dysfunction) at 30, 90 and 365 days and other AKI episodes at one year. In the patients who develop AKI, urinary markers of mitochondrial injury will also be measured at 30 days.

EXPECTED RESULTS:

A 50% reduction in the incidence of AKI in the intervention group compared to the control group is expected. At the same time, markers of mitochondrial damage are expected to be validated in our cohort as biomarkers of AKI progression and to investigate its usefulness as biomarkers of transition to Chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective or urgent heart surgery with extracorporeal circulation at the Hospital Clínic de Barcelona.
* Valve and/or aortocoronary bypass surgery
* Risk of AKI >30% according to the Leicester Cardiosurgery scale

Exclusion Criteria:

* End-stage kidney disease stage V
* Patients with AKI in the 7 days prior to surgery
* Interstitial glomerulonephritis or vasculitis
* Pregnancy
* Kidney transplant
* Endocarditis
* Patients with mechanical assistance devices (ECMO, LVAD, RVAD, IABP)
* Inclusion in another clinical intervention test during the intervention period
* Emergence surgery
* Patients in need of pressure-directed therapy of cerebral infusion.
* Constrictive pericarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
AKI incidence | 18 months
  Reduction in the incidence of AKI

SECONDARY OUTCOMES:
Major kidney adverse events (MAKE) at 30, 90, 365 days | 12 months
  To evaluate the incidence of MAKE in both groups
ICU and hospital length of stay | 18 months
  Days of ICU and Hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Poch, PhD, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No